CLINICAL TRIAL: NCT05766800
Title: Induction Therapy With PD-1 Antibody Combined With Platinum-based Doublet Chemotherapy for Locally-advanced Non-small Cell Lung Cancer: A Randomised Controlled, Open-label, Phase 2 Trial
Brief Title: Induction Therapy With PD-1 Antibody Combined With Platinum-based Doublet Chemotherapy for Locally-advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-013
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; 130-nm albumin-bound paclitaxel; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Downstaged arm with surgical treatment (Experimental): In this arm, patients with tumors resectable after chemoimmunotherapy will receive surgical treatment in department of thoracic surgery.
  Interventions: Drug: Serplulimab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Nab-paclitaxel; Drug: Liposomal paclitaxel; Procedure: Surgery
- Downstaged arm with radiotherapy (Active Comparator): In this arm, patients with tumors resectable after chemoimmunotherapy will receive radiotherapy in department of medical oncology.
  Interventions: Drug: Serplulimab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Nab-paclitaxel; Drug: Liposomal paclitaxel; Radiation: Radiotherapy
- Unresectable arm (Other): In this arm, patients with tumors still unresectable after chemoimmunotherapy will receive therapy in department of medical oncology.
  Interventions: Drug: Serplulimab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Nab-paclitaxel; Drug: Liposomal paclitaxel; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Serplulimab — Specified dose on specified days
Drug: Carboplatin — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Nab-paclitaxel — Specified dose on specified days
Drug: Liposomal paclitaxel — Specified dose on specified days
Procedure: Surgery — Patients with stage IIIB-IIIC non-small cell lung cancer are treated with nab-paclitaxel/pemetrexed plus carboplatin and serplulimab for 4 cycles. Those with downstaged and resectable tumors after chemoimmunotherapy are randomised into surgical treatment arm and radiotherapy arm, and those with tumors still unresectable after chemoimmunotherapy will receive non-surgical treatment in department of medical oncology in the third arm.
  Arms: Downstaged arm with surgical treatment
Radiation: Radiotherapy — Patients with stage IIIB-IIIC non-small cell lung cancer are treated with nab-paclitaxel/pemetrexed plus carboplatin and serplulimab for 4 cycles. Those with downstaged and resectable tumors after chemoimmunotherapy are randomised into surgical treatment arm and radiotherapy arm, and those with tumors still unresectable after chemoimmunotherapy will receive non-surgical treatment in department of medical oncology in the third arm.
  Arms: Downstaged arm with radiotherapy; Unresectable arm

SUMMARY:
For unresectable locally-advanced non-small cell lung cancer, chemoradiotherpay plus immunotherapy is recommended by PACIFIC trial. However, it is unclear whether surgery can provide survival benefit for patients with tumors initially unresectable transformed into resectable ones after chemoimmunotherapy. This trial aims to investigate the efficacy and safety of the therapeutic regimen of chemoimmunotherapy plus surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and stage IIIB-IIIC confirmed by imageological examinations (CT, PET-CT or EBUS).
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.)
8. Patients with normal lung function can tolerate surgery;
9. Without systematic metastasis (including M1a, M1b and M1c);
10. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of Serplulimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
11. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of Serplulimab (whichever is later).

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
4. Participants who are allergic to the test drug or any auxiliary materials;
5. Participants with Interstitial lung disease currently;
6. Participants with active hepatitis B, hepatitis C or HIV;
7. Pregnant or lactating women;
8. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
9. Participated in another therapeutic clinical study;
10. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 30 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 4 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.
Major pathologic response (MPR) | up to 5 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery
Progression-free survival (PFS) | up to 60 months
  It refers to the time (months) from the first administration of drug in this study to the disease progression or death (including any cause of death in the case of no progression) as recorded in CRF, regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.
Disease-free survival (DFS) | up to 60 months
  It refers to the time (months) from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Duration of response (DOR) | up to 60 months
  It is defined as the time from the first time of partial response or complete response to progressive disease via RECIST1.1.
Disease-control rate (DCR) | up to 60 months
  It is defined as the rate of stable disease, partial response, or complete response via RECIST1.1.
R0 rate | up to 5 months
  It is defined as the rate of complete resection with no residual tumor cell in the resection margin.
Severe adverse event (SAE) rate | up to 6 months
  It is defined as the frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.
Health related quality of life (HRQol) | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.